CLINICAL TRIAL: NCT05974384
Title: Music During the Reduction of Distal Radius Fractures as an Adjunctive Therapy for Pain and Anxiety Management: A Randomized Controlled Clinical Trial
Brief Title: Music During the Reduction of Distal Radius Fractures as an Adjunctive Therapy for Pain and Anxiety Management.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Heber Enrique Cueva Sevieri, Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Music Radio
Record Dates: First submitted 2023-07-14; First posted 2023-08-03 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Distal Radius Fracture Reduction
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Music (Placebo Comparator): Intervention without music
  Interventions: Device: No Music
- Music (Active Comparator): Intervention while listening to music
  Interventions: Device: Music

INTERVENTIONS:
Device: No Music — No listening to music while intervention is carried out
  Arms: No Music
Device: Music — Listening to music while intervention is carried out
  Arms: Music

SUMMARY:
Fractures of the distal end of the radius are one of the most frequent fractures diagnosed in the emergency room. The initial management, and in many cases definitive, is carried out through manipulation, closed reduction and immobilization in the emergency room. Different methods of anesthesia have been described to reduce pain during the manipulation and reduction procedure, such as: hematoma block, periosteal block, general anesthesia, intravenous regional anesthesia, nitrous oxide, intramuscular sedation, and conscious sedation. Despite the use of different methods of anesthesia, none is fully effective and each of these methods is not free of complications. Adjuvant measures could play an important role in improving the patient's experience during the procedure, however, there is little evidence in this regard.

Music is increasingly being studied and developed as an adjunctive therapy in the management of pain and anxiety in different medical procedures, demonstrating a statistically significant reduction in pain and anxiety. However, in the literature there is no evidence of studies that evaluate the effect of music during the reduction of fractures in traumatology as an adjuvant therapy for the management of pain and anxiety.

In our experience, despite the anesthesia used, reductions of distal radius fractures are usually a painful procedure that involves a certain degree of discomfort for the patient. For this reason, the investigators believe this study is necessary, as it could demonstrate a new adjuvant therapy that reduces pain and anxiety and improves the overall experience of the patient, in addition to being music, a low-cost tool with no risks for patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Clinical and radiological diagnosis of a fracture of the distal end of a closed radius that has an indication for closed reduction.

Exclusion Criteria:

* Diagnosis of other concomitant fractures.
* Allergy to local anesthetics.
* Significant hearing impairment and/or use of hearing aids.
* Patients whose comorbidities prevent correct participation in the procedure (such as cognitive impairment, diagnosis of psychiatric diseases, patients under the influence of drugs...).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in VAS scale for pain | Will be completed just after the fracture immobilization
  It will be completed after the procedure and the punctuation will go from 0 to 10
Change in Anxiety STAI-6 | Done just before and after the pfracture immobilization
  Puntuation between 20 and 80, 50 considered high anxiety level

SECONDARY OUTCOMES:
Cardiac frequency | Will be assessed just before, during and after the fracture immobilization
  Measurement of the cardiac frequency assessed before, during and after fracture immobilization
Blood pressure | Will be assessed just before, during and after the fracture imobilization
  Measurement of the blood pressure will be assessed before, during and after fracture immobilization
Satisfaction after procedure | Just after the immobilization, when patient will be discharged
  1 to 5 scale for satisfaction with the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chhabra AB, Yildirim B. Adult Distal Radius Fracture Management. J Am Acad Orthop Surg. 2021 Nov 15;29(22):e1105-e1116. doi: 10.5435/JAAOS-D-20-01335. PMID 34288886
- [Background] Tabrizi A, Mirza Tolouei F, Hassani E, Taleb H, Elmi A. Hematoma Block Versus General Anesthesia in Distal Radius Fractures in Patients Over 60 Years in Trauma Emergency. Anesth Pain Med. 2016 Nov 27;7(1):e40619. doi: 10.5812/aapm.40619. eCollection 2017 Feb. PMID 28920036
- [Background] Lee JH. The Effects of Music on Pain: A Meta-Analysis. J Music Ther. 2016 Winter;53(4):430-477. doi: 10.1093/jmt/thw012. Epub 2016 Oct 19. PMID 27760797
- [Background] Sprague S, Scott T, Dodds S, Pogorzelski D, McKay P, Harris AD, Wood A, Thabane L, Bhandari M, Mehta S, Gaski G, Boulton C, Marcano-Fernandez F, Guerra-Farfan E, Hebden J, O'Hara LM, Slobogean GP; PREP-IT Investigators. Cluster identification, selection, and description in cluster randomized crossover trials: the PREP-IT trials. Trials. 2020 Aug 12;21(1):712. doi: 10.1186/s13063-020-04611-9. PMID 32787892
- [Background] Low S, Papay M, Eingartner C. Pain Perception following Initial Closed Reduction in the Preoperative Care of Unstable, Dorsally Displaced Distal Radius Fractures. J Hand Microsurg. 2019 Aug;11(2):111-116. doi: 10.1055/s-0039-1688681. Epub 2019 May 26. PMID 31413496